CLINICAL TRIAL: NCT03653078
Title: Evaluation of Root Proximity During Mini-Screw Insertion Using a Digital Three-Dimensional Printed Guide Versus Conventional Free Hand Placement Technique in Adult Orthodontic Patients A Split Mouth Randomized Clinical Trial
Brief Title: Root Proximity During Mini-Screw Insertion Using a Digital Three-Dimensional Printed Guide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadir Aboshady, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-08-27
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Orthodontic Appliance Complication
Keywords: Surgical guide; Surgical stent; orthodontic mini screw; temporary anchorage device

STUDY DESIGN:
Intervention Model Description: adult orthodontic participants
Who Masked: Participant, Outcomes Assessor
Masking Description: during the insertion procedure the principle investigator and the co supervisor couldn't be blinded, as the two insertion techniques are completely different.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three dimensional printed digital guide (Experimental): one mini-screw will be inserted in the buccal interradicular space between upper second premolar and first molar using Three dimensional printed digital guide, which is a device deisgned and printed through CAD/CAM technology, it's a printed plate fit on the teeth and buccal mucosa with a channel for mini- screw insertion, mini-screw will be inserted through the plate's channel
  Interventions: Device: Three dimensional printed digital guide
- Conventional free hand insertion (No Intervention): one mini-screw will be inserted in the buccal interradicular space between upper second premolar and first molar using conventional free hand insertion of mini-screw, which is a technique using the guiding anatomy for mini-screw insertion using the driver and the operator's skill.

INTERVENTIONS:
Device: Three dimensional printed digital guide — A CAD/CAM printed plate with a channel for mini-screw insertion
  Other Names: surgical guide; surgical stent
  Arms: Three dimensional printed digital guide

SUMMARY:
Although mini screw insertion is considered as a simple and non-invasive technique, it's a critical procedure which requires precision and accuracy. The placement of mini-screw poses a challenge to the orthodontist, particularly if the space available for mini-screws is limited.4 The proximity to the vital structures surrounding the proposed mini-screw position necessitates the precise knowledge of the anatomy of the insertion area.5 The incidence of mini-screw to tooth contact in the placement of inter-radicular region was 27%.6 Although failure of mini screw is considered a multi-factorial concern, many studies reported the proximity of a mini-screw to tooth structures is a major risk factor for failure, especially in the inter-radicular inserted mini-screws. guided insertion was believed to give more favorable results. Above all, the recent technology of the scanning and three-dimensional printing could pave the way to construct a simple accurate guide. Additionally all previous studies assessed the insertion accuracy using CBCT post-operatively, that can't be applied on human subjects for ethical reasons. Thus a non-invasive method for assessment of mini-screw insertion should be implemented.

DETAILED DESCRIPTION:
PICOs P: Adult orthodontic patients need mini screws in maxillary arch bilaterally for anchorage I: Three dimensional printed digital guide for mini screw insertion C: Conventional free hand insertion technique

- O: Primary outcome: Root proximity

Secondary outcomes:

* Patient discomfort during insertion 17
* Insertion accuracy
* Angular deviation
* Linear deviation
* Failure 18 S: Split Mouth Randomized clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic patients with Angle's Class I bimaxillary protrusion • Patients having average mandibular plane angle

Exclusion Criteria:

* Mixed dentition patients

  * Smoker patients
  * Patients with Increased lower facial height
  * Patients with missing posterior teeth
  * Bleeding disorders or anticoagulant therapy
  * Patients with cleft lip & palate
  * Patients with facial asymmetry
  * Patients with transverse maxillary deficiency

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Root proximity | immediately after mini-screw insertion (T0)
  Distance between inserted mini screw and the adjacent roots in microns

SECONDARY OUTCOMES:
Patient discomfort: | immediately after mini-screw insertion (T0)
  Likert scale, it is scale divided into five points to measure the degree of patient discomfort maximum value(5) strongly discomfort, discomfort, neutral, little discomfort, and minimum value (0)no discomfort

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bae MJ, Kim JY, Park JT, Cha JY, Kim HJ, Yu HS, Hwang CJ. Accuracy of miniscrew surgical guides assessed from cone-beam computed tomography and digital models. Am J Orthod Dentofacial Orthop. 2013 Jun;143(6):893-901. doi: 10.1016/j.ajodo.2013.02.018. PMID 23726340
- [Background] Suzuki EY, Suzuki B. Accuracy of miniscrew implant placement with a 3-dimensional surgical guide. J Oral Maxillofac Surg. 2008 Jun;66(6):1245-52. doi: 10.1016/j.joms.2007.08.047. PMID 18486791